CLINICAL TRIAL: NCT04245007
Title: Effect of 8 Weeks 5:2 Intermittent Fasting on Fat Mass Among Obese Male Students Aged 18-25 in Indonesia University
Brief Title: Effect of Intermittent Fasting on Fat Mass
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Hadiyati Fudla, Master Student at Faculty of Medicine, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KET/1354/UN2.F1/ETIK
Record Dates: First submitted 2020-01-18; First posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Obesity
Keywords: obese; intermittent fasting; fat mass; body fat reduction
MeSH Terms: conditions — Obesity; Intermittent Fasting | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Subject will ask to do 5:2 intermittent fasting (2 non-consecutive days a week) within 8 weeks
  Interventions: Behavioral: Fasting
- Control (No Intervention): Subject will prohibited from doing fasting or intake restriction within 8 weeks

INTERVENTIONS:
Behavioral: Fasting — Doing fasting 2 days a week within 8 weeks
  Arms: Intervention

SUMMARY:
This study is aimed to assess the different effect on fat mass between fasting (intervention) group and not fasting (control) group after 8 weeks 5:2 intermittent fasting (IF) among obese male student aged 18-25. Female students are excluded because if they do any restriction intake during their menstruation period which is a lot of blood lost, it will be a risk for them.

This study is designed as non-blinding randomized control trial. Subject who adhere with less than 85 percent fasting (14 out of 16) will be dropped out from this study. Total sample in this study is 62 students which are 31 students for each group.

DETAILED DESCRIPTION:
5:2 intermittent fasting (IF) is eating pattern in which no or few calories are consumed for 13 hours (for 5 am to 6 pm) done in two non-consecutive days days per week, followed by ad libitum intake on the remaining days, without any requirement of water restriction.

Subjects will be distributed to each group by using randomization block of four.

This study will use 8 forms consist of; informed consent, subject selection form, re-anthropometric measurement form, questionnaire, semi quantitative food frequency questionnaire (SQ-FFQ), international physical activity questionnaire (IPAQ), food record book, and control and evaluation form. While the tolls are consist of food photograph book (to help in filling the food record book), body height scale, and bio-electrical impedance analysis (BIA) Seca medical body composition analyzer (mBCA) 515/514 (to measure body composition).

ELIGIBILITY:
Inclusion Criteria:

* obese male student age 18-25
* do not have experience on amputation
* willingness to participate in the whole study by signing informed consent

Exclusion Criteria:

* hypertrophy muscle students identified from body composition measurement
* in a certain diet at the moment
* consuming lipid-lowering drug at the moment
* doing regular fasting (2 days a week) for 2 months before the study begin
* suffer from chronic illness (confirmed by disease history form
* using electronic implants, for example pacemaker or pane
* using prostheses (artificial body part)

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2020-01-27 (Estimated); Primary Completion 2020-04-09 (Estimated); Study Completion 2020-04-09 (Estimated)

PRIMARY OUTCOMES:
Fat mass | 8 weeks
  reduction fat mass in the intervention group measured by bio-electrical impedance analysis

CONTACTS AND LOCATIONS:
Overall Officials: Hadiyati HF Fudla, Principal Investigator — Indonesia University
Locations (1):
- Indonesia University, Depok, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No